CLINICAL TRIAL: NCT00707005
Title: Antibiotic Susceptibility of Conjunctival Bacterial Isolates From Refractive Surgery Patients
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Kyoung Yul Seo M.D., Yonsei University Health System
Other Study IDs: 4-2008-0164
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Bacterial Keratitis
Keywords: antibiotic susceptibility; bacterial flora; fluoroquinolone; LASIK; refractive surgery

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Conjunctival swab samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the in vitro antibiotic susceptibility patterns of conjunctival bacterial flora isolated preoperatively from patients undergoing refractive surgery.

DETAILED DESCRIPTION:
Laser in situ keratomileusis (LASIK) is the most commonly performed refractive surgical procedure for the correction of ametropia worldwide. Infectious keratitis, although rare, is a potentially devastating complication of LASIK, and it can lead to horrifying outcomes. Previous studies on antibiotic susceptibility of preoperative ocular bacterial flora focused primarily on intraocular surgeries with particular interests in endophthalmitis. This study was aimed at refractive surgeries with special interest in infectious keratitis after LASIK. Intraocular surgeries for cataract, glaucoma or retinal disease are performed mostly on aged patients at a large hospital on an inpatient or outpatient basis; however, most refractive surgeries are performed on young, healthy people in private clinics on an outpatient basis. The patient populations are therefore quite different between these two types of surgery. The aim of this study is to determine the in vitro antibiotic susceptibility patterns of conjunctival bacterial flora isolated preoperatively from patients undergoing refractive surgery at an outpatient laser surgery clinic. Preoperative conjunctival swab samples are directly inoculated in culture media at the bedside before topical anesthetic or antibiotic application. Blood agar, chocolate agar, thioglycolate broth, Sabouraud dextrose agar, and Ogawa media are used for bacterial, fungal and mycobacterial cultures. Minimum inhibitory concentrations (MICs) of ofloxacin (OFX), levofloxacin (LEV), gatifloxacin (GAT), moxifloxacin (MOX), gemifloxacin (GEM) and other commonly used antibiotics are determined using an E-test.

ELIGIBILITY:
Inclusion Criteria:

* Myopia patients scheduled for refractive surgery

Exclusion Criteria:

* Active keratitis
* Current treatment of antibiotics (systemic or topical)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Myopia patients scheduled for refractive surgery
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Minimum inhibitory concentrations of commonly used antibiotics are determined using an E-test. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Yul Seo, M.D., Study Chair — Yonsei University
Locations (1):
- Yonsei University Health System, Seoul, Kyoungkido, South Korea

REFERENCES:
- [Background] Mino de Kaspar H, Koss MJ, He L, Blumenkranz MS, Ta CN. Antibiotic susceptibility of preoperative normal conjunctival bacteria. Am J Ophthalmol. 2005 Apr;139(4):730-3. doi: 10.1016/j.ajo.2004.10.007. PMID 15808182